CLINICAL TRIAL: NCT00173069
Title: A Study on Psychopathological Progress of Early Schizophrenia-Like Disorder (SOPRES)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700403
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; PPI; P50I; MRS; Niacin; Candidate Genes
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This PPG entitled "A Study on Psychopathological Progress of Early Schizophrenia-like Disorder (SOPRES)" is designed to study the "Progress of Psychopathology" of pre-psychotic state of schizophrenia (SCH) using a prospective follow-up design. Based on the neurodevelopment hypothesis of schizophrenia, the neurobiological dysfunctions, such as cognitive impairment, neurophysiological dysfunction, neuroanatomical pathology, is the core pathology. The pathology may exist prior to onset of psychotic symptoms, and at post psychotic state. It also presents in the first-degree relatives. SCH is mainly with a gradual mode of onset, ranging from pre-schizotypal (or pan-neurotic state), schizotypal, prodromal to frank psychotic SCH (DSM-IV criteria) state.

Up to the present time, there are arbitray criteria for diagnosing schizotypal disorder and frank psychiatric schizophrenia, but the valid clinical assessment method of pre-schizotypal and prodromal state is still controversial. The psychopathological progress from pre-schizotypal to frank psychotic SCH state is still unclear. In this SOPRES, we intend to establish a set of valid clinical assessments for defining the cases of early SCH-like disorder [ESLD], to examine the clinical progression, such as conversion rate of psychosis from non-psychotic state in a prospective longitudinal follow-up; to validate the clinically defined cases of ESLD with different dimensions of neurobiological studies, including niacin skin flush test, neuropsychological, neurophysiological (such as prepulse inhibition [PPI], P50 inhibition [P50I]), and magnetic resonance spectrometry (MRS) and Diffusion Tensor Imaging (TDI); to demonstrate the validity of the ESLD using the family genetic-epidemiological data and to explore the awareness, reaction, coping strategy, social stigma, and help seeking process of the patients and the families of ESLD.

In order to achieve these goals, we designed this PPG of SOPRES, which comprises of 4 inter-locked projects and one core unit. Project No.1 is the "Clinical Phenomenological Follow-up Study of ELSD: Clinical Validity"; Project No. 2 is the "Validity Study of Neurobiological Tests of ELSD"; Project No. 3 is the "Validity Study of Family Genetic Study of ELSD"; and Project No. 4 is the "Awareness and Pathways of Help Seeking of ELSD". The only one core unit is designed for the purposed of monitoring research progress, communication among researchers such managing PPG research meeting, data management, and budget management and other research-related administrative secretary work. These 4 projects are integrated study approaches by means of (1) using the same samples; (2) study different levels of psychopathology, including clinical symptoms, neurobiological impairment, family genetic data, and psychosocial variables; and (3) mutual hypothesis testing.

We expect that this SOPRES research will create a new frontier of SCH research in the fields of early intervention of SCH for preventing the recurrence of frank psychotic state of schizophrenia, and will provide the background for improving treatment outcome and quality of life of SCH.

DETAILED DESCRIPTION:
Project No: 1 Title: A Study of Psychopathological Progress of Early Schizophrenia-like Disorder specific aims are 1) To elicit the psychopathology of identified Early Schizophrenia-like Disorder (ESLD) and to categorize into 3 groups of pre-schizotypal, schizotypal, and prodromal ESLD. 2) The reveal the prevalence of different neurobiological impairment (studied in Project No.2) in 3 groups of these identified ESLD subjects. 3) The stability of psychopathology of 3 groups of identified ESLD. 4) The process of conversion and conversion rates of psychotic state from non-psychotic state in a 2-year follow-up

Study procedures:

1. Recruitment:

   The high-risk group of schizophrenia will be recruited by referral from psychiatric outpatient clinics in Northern Taiwan, referral from school counseling room in Taipei City and Taipei County, and subjects with known family history from our previous schizophrenia genetic study, which has a size of 850 families. As we have good collaborative works with several psychiatric hospitals and psychiatric departments of general hospitals, it is expected that 100 subjects could be assessed from the outpatient referral. The increasing needs of psychiatric consultation from school system give us a chance to recruit 50 subjects by school referral (school counseling system). Our previous family genetic studies in schizophrenia have already recruited 850 families. As the relatively risk of schizophrenic spectrum disorders (schizophrenia and schizotypal disorder) is much higher in families with schizophrenic patients, and in our experiences the families of schizophrenic patients often expressed worries about developing the illness themselves, it is expected that 100 subjects could be assessed from this population.

   The school surveillance will be conducted in three selected senior high schools and three colleges in Taipei metropolitan aiming at subjects fitting our recruiting indicators, including cognitive decline, affective symptoms, social isolation, and school failure (CASIS). A pilot study will be conducted in initial 5-10 nominated candidate students to cross check the validity and applicability of each screening methods. There are 75,084 senior high school students in Academic Year 2003-2004 in Taipei City. We plan to survey the teachers of 3000 students to from 3 senior high schools (around 1000 students each), representing schools with highly-academic-, vocational-, and mixed-orientation. Another 3000 students will be recruited from 3 colleges by administering freshman self-report questionnaire. It is expected that 100 subjects could be identified as subjects with early schizophrenia-like clinical presentations.

   The general public will be recruited by respondents to our study ads co-sponsored by the Mental Health Foundation (MHF) framed in terms of highlighting awareness of early cognitive deficits and prevention from severe mental disorders (Caring Brain and Worry Free Program). As the PI had recruited subjects for "brain bank" by public advocacy and the Mental Health Foundation already had annual surveys regarding the general public's mental health conditions and subjective well-being with good response rate and the results have been broadcast on major media. Based on the highly expected credit of the MHF, we expect to identify and recruit 50 subjects from this channel.

   The normal control will be recruited from the subjects' schoolmates or friends not meeting our recruitment criteria, matched by age, gender, and education. We need 200 normal control subjects based on a two to one ration between the study subject and the normal control.
2. Referral criteria:

Outpatient group: suspected "latent" or "beginning of" schizophrenia based on psychiatrists' clinical experiences; school referral group: problematic students unable to be explained by common conduct problems or psychosocial issues from teachers' perspectives (un-understandable emotional, behavioral, interpersonal, or academic problems); family study group: siblings or offspring of schizophrenic patients exhibiting symptoms or behavioral patterns warrant family's attention (something reminding them about their schizophrenic relatives).

3) Recruitment criteria: (CASIS) Cognitive deficits: subjectively poor concentration; decline of intelligence; inefficient learning; rigid thinking; Affective symptoms: unexplainable depressiveness, anxiousness, fearfulness, obsession, or hypochondriacal ideas; social isolation: having less than two close friends; generally withdrew, distant, aloof, or isolated; frequent absence without identifiable causes; school failure: markedly deterioration of academic performance or quitting school.

Subjects presenting at least two of the above conditions (one of cognitive deficit and at least one of the remaining three) will be screened for psychotic-prone symptoms by the Latent Schizophrenia Screening Sheet (LSSS) (necessary to have cognitive deficit) of 26 items (6 dimensions) including thoughts, perceptions, inappropriate behaviors, affective symptoms, interpersonal relationship, and neurotic symptoms. Subjects respond "sure" for any item of the LSS will be recruited for further assessments.

Anticipated Results: The cross-sectional and longitudinal progress of psychopathology of ESLD will be revealed. The comprehensiveness and the domains of psychopathology of ESLD will be elicited. The progressing process of the psychopathological domains will be characterized.

1. The validity of subgrouping of ESLD into pre-schizotypal, schizotypal and prodromal types will be determined.
2. We'll reveal the pattern of aggravation of symptomatic level as time goes by: more subjects progress to the severer level during the 2-year follow-up (i.e., from pre-schizotypy to schizotypy, from prodrome to SCH, etc; few subjects could "drift back" to the milder symptomatic level (i.e., from prodrome to schizotypy or from schizotypy to pre-schizotypy, etc).
3. To determine some specific items in the screening tools, i.e., LSS, SOPS, for better positive predictive values than the others.
4. The sensitivity and specificity of the screening tools will be examined using neurobiological indicators (Project No.2) by constrast validity testing.

Project No: 2 Title: Neurobiological Study of Early Schizophrenia-like Disorder (ESLD) Specific Aims: Based on the neurodevelopmental hypothesis of schizophrenia (SCH), it is assumed that clinically identified pre-psychotic state of SCH, termed as Early Schizophrenia-like Disorder (ESLD)(Project No.1), may have impaired neurobiological functions. Our previous family-based studies also supported that some neurobiological markers, such as sustained attention deficits, were potential endophenotypes of schizophrenia (see background below). Therefore, in Project No.2 of the Study on Psychopathological Progress of ESLD (SOPRES) Program, we plan to adopt multi-level approaches to investigate the potential neurobiological changes in patients with ESLD. The approaches include certain specific neuropsychological, neurophysiological and neuroimaging measurements.

The specific aims of neuropsychological study are as follows: 1) to examine whether individuals with ESLD evidence controlled processing dysfunction of neurocognition; 2) if true, to further explore whether such dysfunction involving neurocognitive domain is simplex or multiplex in nature; 3) to determine whether neurocognitive controlled processing measure(s) used in the present study can be a useful screening tool for ESLD and further for early detection of schizophrenia.

The specific aims of the other dimensions of neurobiological studies are:

1. To clarify the prevalence of impaired flush response to Niacin skin patch in ESLD and to assess the predictive validity of Niacin skin test in the progression of schizophrenia;
2. To reveal the prevalence of two brain inhibitory functions (i.e. prepulse inhibition of startle (PPI) and P50 event-related potential (ERP) suppression) in ESLD and the change along clinical course of those ESLD subjects;
3. To measure the regional changes of magnetic resonance spectroscopy (MRS) in hippocampus and frontal lobe in subjects with ESLD, and define the predictive validity in the follow-up course.
4. To measure the connectivity and diffusion anisotropy between the hippocampus and frontal lobe by diffusion tensor imaging (DTI) in subjects with ESLD, and define the predictive validity in the follow-up course.
5. To evaluate the possibility of skin niacin response/MRS/DTI/P50/PPI as endophenotypes in further genetic research of schizophrenia.

The importance of the specific inhibitory measures also resides in the fact that they are understood at neurobiological (and in some cases, molecular) levels, based on extensive human and animal model studies.

1. P50 Suppression:

   P50 suppression is an important endophenotype of schizophrenia. P50 suppression occurs when two clicks are presented with a 500 msec interstimulus interval. The impaired suppression of the P50 to the second stimulus has been reported in a number of studies in chronic schizophrenia patients, both medicated and unmedicated, first-episode patients, and first-degree relatives of schizophrenics, as well as schizotypal individuals.

   Impaired P50 suppression is extensively studied using anatomical and molecular genetic and other neurobiological studies. These findings support that P50 suppression impairment is a possible endophenotype of information processing deficits in schizophrenia.
2. Prepulse inhibition (PPI):

PPI of the startle response is an operational measure of preattentive sensorimotor gating. The term startle modification refers to the changes in the startle reflex, induced by various stimulus modalities, when the startle-eliciting stimulus is preceeded by a (usually weak) stimulus called a prepulse. It is stable over time in both normal subjects and schizophrenia patients.

Deficits in PPI have been consistently identified in schizophrenia, and PPI is an excellent candidate endophenotype in schizophrenia since PPI deficits occurred in schizophrenia patients, and schizotypal personality disorder patients.

To study the presence and change of impaired PPI and P50 suppression in ESLD may help us clarify the stability of the impairment along the disease course and the validity of using the PPI and P50 test as a screening tool for pre-psychotic state of schizophrenia.

Project No: 3 Title: Family Genetic Study of Early Schizophrenia-like Disorder I. Specific Aims: Genetic high-risk (HR) approach, in which subjects with one or more affected relatives were recruited since infancy or early childhood, has been the most commonly adopted one to address the early detection of schizophrenia (1). However, as pointed out in a recent review (2), there are two major limitations of these studies. First, because the majority of these genetic high-risk studies were started 30-40 years ago, many of them used methods that are outdated and sometimes focused on less relevant subjects in their assessments. Second, only approximately 10% of the HR children develop schizophrenia, making the predictions concerning vulnerability indicators unprecise. Recently an alternative approach called clinical high-risk or ultra-high-risk has been advocated, in which adolescents or young adults referred for mental health evaluation with attenuated psychotic symptoms or behavioral problems commonly observed in the HR children were recruited for prospective follow-ups (3, 4). In this PPG, we propose an approach that combines both genetic HR and clinical HR to enrich the recruitment of subjects at increased risk of developing early schizophrenia-like disorder (ESLD).

Moreover, the interpretation of the contrast between HR subjects and normal controls or between HR with onset of schizophrenia and HR without onset of schizophrenia tends not to be straightforward. Any neurodevelopmental disturbances can be distributed in two independent dimensions: a genetic-environmental causal continuum and an early-to-late maturation expression continuum (5). A factor that is present in an HR subject but absent in normal controls is not necessarily of genetic origin. One way to distinguish is to examine whether a similar deficit is present in other non-HR sibling of the HR proband. However, previous HR studies tended to measure only the HR subject in each family.

In this component project, we propose to adopt a family-genetic approach to provide more information for the interpretation of the contrast between HR of different severity and normal controls or between HR with progression to a more severe stage and HR without such progression. The specific aims of this component project are as follows:

Aim 1:To assess to what extent the psychopathological features identified in the probands of pre-schizotypal ESLD, schizotypal ESLD, prodromal ESLD, or early schizophrenia are also present in their first-degree relatives.

Aim 2: To assess to what extent the neurodevelopmental or neurobiological impairment identified in the probands of pre-schizotypal ESLD, schizotypal ESLD, prodromal ESLD, or early schizophrenia are also present in their first-degree relatives.

Aim 3: To assess to what extent the conversion in psychotic-like state of the three groups of ESLD probands can be explained by the presence of psychopathological, neurodevelopmental, or neurobiological features observed in their first-degree relatives.

The probands of the three groups of ESLD (pre-schizotypal ESLD, schizotypal ESLD, and prodromal ESLD), early schizophrenia, and normal controls will be recruited by the Component Project 1 of this PPG. On the basis of these probands, this Component Project will recruit their first-degree relatives to participate in the study. Part of these probands will have neurobiological assessment conducted in Component Project 2. Part of the family identified in this Component Project will be evaluated for help-seeking behavior. In these joined efforts, we will be able to decipher the psychopathological pathways for both genetic and environmental etiological factors.

Core Unit Code No: A Title: Core Unit of A Study on Psychopathological Progress of Early Schizophrenia-like Disorder (CUSOPRES) This PPG of Study on Psychopathological Progress of Early Schizophrenia-like Disorder (ESLD) [SOPRES] is composed of 4 inter-related projects: (1) A Phenomenological Prospective Follow-up Study of ESLD; (2) A Neurobiological Study of ESLD; (3) Family Genetic Study of ESLD; (4) Awareness and Pathways to Care in ESLD.

The study samples participate all these four projects. The major hypothesis of the SOPRES was based on neurodevelopmental etiological hypothesis of schizophrenia. The hypothesis testing is interrelated among three projects No.1, No.2 and No.3. The projects No.4 is supplementary to other 3 projects. This SOPRES belongs to a translational study. Project No.4 is essential to bridge the process for clinical application of this SOPRES.

Based on these predicted research activities commonly needed for these four projects of this PPG, an efficient Core Unit of this SOPRES (CUSOPRES) is mandatory for carrying out the research work smoothly. There are several sections of research-related work of this CUSOPRES

1. Administrative Coordination of this SOPRES:

This CUSOPRES has to coordinate the regular research meeting, to make record of this research meeting. Literature related to this SOPRES PPG has to be collected and to be distributed to all research participants. It has to monitor the reality of the progress of this SOPRES. The progress of sampling, data collection, data check, setting up computer data file has to be monitored weekly. Report of research progress has to be done and has to be distributed to all main researchers. All the filing system of this SOPRES has also to be done by this CUSOPRES.

2. Budget management: Some proportion of the budget are commonly used in three projects. Each project also has its own budget schedule. The salary system of all research assistant has to be scheduled and managed clearly. This budget is of government grant. Detailed descriptions and records of budget expenditure are critically demanded by the regulatory and census system of the government. The expenditure every year must to be regulated to meet the requirement of research activity. This CUSOPRES has to manage all these works. A full time business assistant is necessary.

3. Training of Research Assistants and Participant Researchers: This PPG OF SOPRES will recruit research assistants (RA) for sampling, for data collection and data management. In Taiwan, the job of RA is always in a temporary basis. They (RA) come and go. All these RA's enrolled have to receive a through training for their work to guarantee high training of data collection and data management. All participant young researchers of all different disciplines also have to arrange training program related to the SOPRES research activities. This training program has to be arranged, scheduled and managed by the CUSOPRES.

4. Manuscript Preparation and Submission. Other than collecting new data, this PPG also have abundant data bank of previous psychopathological studies. As stated in the preliminary work of these three projects, these data has to be analyzed along the progress of data collection of this SOPRES. These continuous data analysis will create many drafts of paper manuscripts. Thus, this SOPRES PPG will have many manuscripts preparations for submitting to international and/or domestic journals. Typing, editing, and the preparation of these manuscripts are part of the work of this CUSOPRES. This is one important supporting function of CUSOPRES.

5. Data management and Data Analysis After preliminary management of data collected from the study subjects, all research data have to be set up in suitable computer data bank. Data cleaning is important work. Integrated data analyses of this SOPRES are unique of this SOPRES PPG. Other than independent analysis of the specific project itself, coordinated and mutual data matching analysis is unique of this SOPRES. The clinical definition of ESLD will be validated by concurrent psychopathological data (Project No.1) and follow-up data, and will be validated by all different dimensions of neurobiological data (Project No.2). The clinically defined ESLD will also be validated by family genetic data. Most importantly, heterogeneity of ESLD will also be explored using statistical maneuvers and then, will receive further validation study.

Data Structure and Statistical data analysis

Figure1 illustrates the possible data relationship and statistical analysis tools and data analysis strategies to be involved in and incorporated into the project. Structure of data sets to be collected by four component projects is very complicate in nature:

1. . Data sets to be collected by all four projects are inter-correlated and dependent. Subjects may be stratified by various relationships among all four projects.
2. . Data sets are highly multidimensional. Each program project employees multiple interviewing and measurement tables. Subjects match different criteria may have different sets of measurements.
3. . These measurements have different scales: ratio, interval, ordinal, nominal. Multivariate variables with different scales will be studied simultaneously.
4. . Some of the subjects/measurements combinations may have longitudinal pattern with follow-up studies.
5. . Data sets collected by Project 3 may be of dependent nature - samples are clustered as families.

Due to the high complexity of the data structure involved, the core unit has the following strategies to handle the statistical data analyses for all different project/subject/table/variable combination and situation:

1. . Descriptive statistics and various exploratory data analysis (EDA) tools will first be used to study the basic distribution structure for all the subjects/variables collected. This provides the researchers most of the univariate distributions and some of the associations structure of tables.
2. . Generalized association plots (GAP), developed by Dr. Chun-houh Chen (Chen 2002) for our previous projects, will also be used to explore the basic clustering structure of subjects and grouping structure of variables and the interaction patterns of the subject-clusters with variable-groups for each individual data table and combination of tables. This provides us an overall picture of data structure for all the subjects/tables involved.
3. . Many conventional multivariate statistical analysis tools will be employed to conduct further exploratory analyses and some confirmatory studies for the data.
4. . Various statistical testing procedures will also be used to verify and answer some of the hypotheses generated and proposed by all four component projects. The results may lead to new or modified hypotheses. Statistical analyses and hypothesis testing procedures will be performed again to verify the new hypotheses.
5. . Various statistical and epidemiological genetic analysis tools are to be used for analyzing the familial data generated by project 3.
6. . Latent class model (LCM) developed by Dr. Huang (Huang & Bandeen-Roche 2004, Huang 2005) can be used to study subject clustering pattern for various project/table combination.
7. . CateGAP, longGAP, canoGAP will be applied to study the categorical, longitudinal, and canonical relationship data structure respectively.
8. . New statistical methodologies and data analysis procedures suitable for analyzing specific data pattern to be generated by all four projects will be developed by the statisticians of the core unit when there is the need.

6. International and Domestic Communication Related to academic activities of this SOPRES, this SOPRES focuses on the up-to-date psychopathological study issue. All participant researchers of this SOPRES have abundant communication with other academic institutes or personnel for academic interests. This CUSOPRES has to manage all these communications.

7. The GENOP research team of this SOPRES program has also done the positional cloning study in order to find the vulnerability gene of schizophrenia in an independent molecular genetic study on SCH. We have found 12 potential candidate vulnerability genes up to now. In the coming years, there will be risk mutations identified in these vulnerability genes. These risk mutations will be as the direct genetic marker to validate the different groups of ESLD. This core unit will hire one assistant of bachelor degree to do blood sample collection and DNA extraction, as well as lymphocyte immortalization by EBV transformation.

8. Summary and Significance

This PPG of "A Study on Psychopathological Progress of Early Schizophrenia-like Disorder (SOPRES)" was designed to validate Early Schizophrenia-like Disorder (ESLD) defined clinically, using neurodevelopmental-associated core psychopathology. The SOPRES will recruit subjects of potential cases of ESLD using clinical psychopathological data obtained by self-report and face-to-face interview approach. Three groups of ESLD will be defined: (1) pre-schizotypal (or pan-neurotic), (2) schizotypal and (3) prodromal groups. These three groups represent three steps of psychopathological progress of ESLD. Using prospective follow-up design, the conversion rates of these three groups converted into successive group and into frank psychotic state of schizophrenia will be revealed. These clinically defined cases will be validated using neurobiological indicators, such as neuropsychological, neurophysiological, niacin skin flushing test, neurochemical, neuroanatomical indicators (Project No.2) as well as family genetic epidemiological data (Project No.3). The subtypes of ESLD will also be delineated using these validation procedures. The awareness, reaction and coping strategy of the patients and the family care-givers will be elicited as well. This SOPRES is 5-year study design, which includes 4 study periods: (1) half year preparation, (2) 2 years of case recruitment, (3) 2 years of follow-up and (4) half year ending and data management.

The psychopathology of schizophrenia has been well studied in the past decade. The SOPRES is a translational study design to examine the psychopathological progress of the pre-psychotic state of schizophrenia based on neurodevelopmental hypothesis of schizophrenia. This SOPRES is, thus, of high academic merit in the study of schizophrenia psychopathology. This SOPRES will demonstrate the successful application of basic neurobiological study data on clinical condition of ESLD.

This SOPRES will successfully set up a battery for valid diagnostic assessment of ESLD covering multidimensional psychopathology and it will also reveal the psychological progress of ESLD. This valid diagnostic assessment of ESLD will identify cases of ESLD from the cases with school failure, job difficulty, and of anxiety-depressive disorders in general psychiatric clinics. This will be helpful for avoiding the undesirable clinical condition of mis-diagnosis and mis-treatment. This will also substantiate the background for the development of further frontier of early intervention of ESLD. As schizophrenia is a devastating disease for the patient himself/herself, the family and the society. It also carries heavy psychosocial stigma. The result of SOPRES will be very helpful for building up early, intervention of schizophrenia, and will contribute a lot in reducing the cost of schizophrenia. The SOPRES study results regarding the awareness and coping strategy of the patients and the family will provide useful empirical data for developing psychosocial service for the ESLD.

This SOPRES study will provide the learning experience for participating researchers, including research assistants in the area of developing diagnostic assessment, combing clinical psychopathology and neurobiological pathology of early pre-psychotic state of schizophrenia. This experience will cultivate the future professional persons in the research area of preventive psychiatry.

9. Institutional Environment and Resources

This PPG of SOPRES will be carried out with the main researcher center located at the Department of Psychiatry, National Taiwan University Hospital and College of Medicine, National Taiwan University. There are main psychiatric hospitals affiliated with this research center. Massive case and family recruitment in local and nationwide programs for molecular genetic study of schizophrenia has been carried out by this research center and the affiliated hospitals. This research center has been doing psychopathological study on schizophrenia in its academic tradition. This research center is one part of the active medical campus of the National Taiwan University. Multidisciplinary team related to neurobiological study has been organized for years. These neurobiological studies of neuropsychological, neurophysiological and neuroimaging fields and neurobiological technology have been well developed. This university medical campus is very active in collaborating with other research sections as shown by this PPG of SOPRES. The Department of Imaging, Department of Neurology, Department of Nursing, and Department of Psychiatry, College of Medicine; Department of Psychology, College of Science, Department of Social Worker, College of Social Science, Institute of Epidemiology, College of Public Health of the same University are integrated with this PPG. The active research centers of statistical science located in Academia Sinica, and National Chiao Tung University, as well as Institute of Anthropology, National Tsing Hua University are also integrated into this PPG of SOPRES. These institutions are all engaged in biomedical research actively and also encouraging researchers to pursuit incultidisciplinary collaborative research too. The clinical phenomenological study, follow-up study, genetic laboratory, the neuropsychological, neurophysiological, the neuroimaging technique, and statistical technology are well equipped and well developed in these collaborative research centers and well mastered by these participating researchers.

Besides, this research center is the leading center of psychopathological study and service in the area of adolescent Psychiatry. There was wide and intensive connection between this research center and schools. Besides, this research center has also been involved with public mental health promotion through Mental Health Foundation (MHF). These intensive connections and wide resources are crucial for the successful case recruitment of ESLD targeted by this SOPRES program.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* one or two schizophrenia sib-paired children, one schizophrenia patient parent and the other one should be normal

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324
Dates: Start 2006-01; Study Completion 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University